CLINICAL TRIAL: NCT07273045
Title: reGISTry - a Comprehensive, Multinational GIST Registry
Brief Title: A Comprehensive, Multinational GIST Registry
Acronym: reGISTTry
Status: Not yet recruiting | Type: Observational
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Johanna Falkenhorst, MD, Universität Duisburg-Essen
Other Study IDs: reGISTTry
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Gastrointenstinal Stromal Tumor (GIST); GIST - Gastrointestinal Stromal Tumor
Keywords: GIST; KIT; SDH-Deficiency; NF1; register
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — During clinical routine procedures, in indicated
  * Blood
  * Tumor
  * Saliva
  * Stool
  * Urine
  * Liquor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all patients with GIST regardless of disease status or molecular subtype

SUMMARY:
Patients diagnosed with a gastrointestinal stromal tumor (GIST), a rare type of tumor in the digestive tractparticipate in this scientific research study, known as a registry study, to help improve understanding and treatment of GIST.

This study collects medical information and biological samples-such as blood or tumor tissue-from patients. It does not involve new treatments, medications, or medical procedures. The patient's regular medical care will continue as usual, and participation will not require extra appointments or tests.

The study aims to learn more about how GIST behaves, especially in rare forms such as SDH-deficient or NF1-associated tumors. While targeted drugs are available for many patients, some tumors return or become resistant to treatment. By gathering data from many patients, researchers hope to better understand these challenges, identify risk factors for worse outcomes, and help design future studies and treatments-especially for rare types of GIST.

If the patient agrees to participate, information will be collected from their medical records, scans (such as CT or MRI), and doctor visits. They may be asked to complete optional questionnaires about their health and quality of life. If they consent, small blood samples (up to 50 ml) may be collected during routine check-ups. If surgery is needed, a small part of the tumor tissue may be stored for research. Other samples-such as saliva, stool, urine, or spinal fluid-may also be collected if they are taken during normal care, to study how bacteria in the body might affect the disease and treatment.

Participation is completely voluntary. The patient can choose to join or not, and can withdraw at any time without affecting their care or relationship with their doctor. Even if they do not agree to provide biological samples, they can still take part in the study by sharing medical data and scan results.

DETAILED DESCRIPTION:
This is a prospective, multi-center observational study aiming to collect clinical data from GIST patients and to longitudinally store radiological and pathological material. Additionally, anonymized retrospective data from the period 1995 to 2025 will be supplemented from existing institutional GIST databases. The study does not currently aim to change current clinical practice in treating GIST patients. Instead, it seeks to generate a robust and consistent dataset to capture oncological outcomes, as well as other outcomes that may improve the quality of care (e.g., surgical results, patient and disease-related risk factors, healthcare research), ultimately enhancing the treatment and counseling of GIST patients.

Patients diagnosed with GIST who meet the inclusion criteria are invited to participate in the current study. Eligible patients receive comprehensive information about the proposed treatment, as well as details on the data and materials (clinical, radiological, and pathological) that will be collected. They are informed that participation will not affect their current treatment. Suitable and informed patients who provide consent are enrolled in the prospective cohort study (PCS) and followed prospectively.

For patients who voluntarily consent to sample collection through the West German Biobank Essen or the externa biobank of üparticipating centers, additional blood samples are collected during planned CT scans of the chest and abdomen-alongside routine blood draws-for storage in the biobank. Patients are also invited to complete optional questionnaires about their quality of life. If a tumor resection is performed, tumor tissue may be stored for research purposes upon consent. If patients choose to continue treatment or follow-up at another center, they may be contacted by phone at regular intervals after giving consent, and asked to complete quality-of-life questionnaires. They may also be asked to share imaging data and medical reports. With consent, the study team will contact the treating physicians to obtain updates on the patient's disease course.

A data collection form has been developed in the REDCap platform at the Institute for Artificial Intelligence in Medicine (IKIM), Essen, Germany. It includes patient- and tumor-related factors, treatment variables, follow-up findings, time to local recurrence, and follow-up status. All participating centers use this shared platform. Retrospective data are stored anonymously, while prospective data are stored pseudonymously. Only the overall study leadership has access to all data.

Each participating reference center can access imaging data (CT or MRI scans) and pathological material (a representative formalin-fixed tumor block) from their own patients. Patient identifiers are removed to ensure confidentiality. All data shared between institutions are de-identified and pseudonymized, and all measures to conceal patient identities are taken. Radiological images are also pseudonymized and stored in the REDCap database. Pathological materials are stored in a decentralized manner within the biobanks of the participating centers. Consent to participate in the biobank is optional.

After a subproject is submitted and approved, pseudonymized data are made available to the respective centers. Each center is responsible for entering and storing its own patient data, imaging results, and pathological samples. At the time of analysis, each center is required to provide updated data upon request.

Personal data are retained only for as long as necessary for study purposes. Data will be deleted no later than 30 years after enrollment. Personal data are only shared with third parties if consent has been given or if a law permits such sharing.

Within the GISTT Research Consortium, anonymized data may be shared upon request with participating centers in Germany and abroad (within and outside Europe), provided a project proposal has been submitted to the overall study leadership and the research question is deemed meaningful and feasible. It is expected that additional centers will join the study over time. All participating centers may submit project proposals. These centers are typically research-focused sarcoma centers at university hospitals worldwide. Data are shared exclusively in pseudonymized form. The distribution of biological samples is also coordinated through the overall study leadership.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a gastrointestinal stromal tumor (GIST)
* Verbal and written informed consent for participation in the study with planned prospective data collection
* Physical and mental ability to provide informed consent

Exclusion Criteria:

* Severe neurological or psychological illness that impairs the ability to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age group with a diagnosis of gastrointestinal stromal tumor (GIST).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2056-01-01 (Estimated); Study Completion 2056-01-01 (Estimated)

PRIMARY OUTCOMES:
Creation of a prospective and retrospective, multi-center, international GIST cohort as a foundation for analyzing prognostic factors and planning future clinical trials. | 30 years

SECONDARY OUTCOMES:
Establishment of a comprehensive biobank with corresponding clinical, radiological, and histological data to support future research projects. | 30 years
Identification of risk factors relevant to the treatment and counseling of GIST patients. | 30 years
Identification of predictive factors for response to local and systemic therapies. | 30 years
Characterization of resistance mechanisms. | 30 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essem, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Ethical Vote Pending